CLINICAL TRIAL: NCT05071001
Title: Long Term Brain Toxicity of Chemotherapy in Patients Treated for a Bone TumorDuring Childhood or Adolescence
Acronym: OSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A00919-30
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Adults Treated During Childhood or Adolescence for a Malignant Bone Tumor (Osteosarcoma and Ewing Sarcoma)
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental)
  Interventions: Procedure: MRI
- B (Experimental)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — This assessment will be planned in the year after the consent signAll patients will have one brain MRI performed in Henri Mondor Hospital on a 3T MR unit (Skyra, Siemens, Erlangen). The procedure will include:
  1. a 3D-FLAIR imaging
  2. a morphometric study based on a 3DT1 MPRAGE gradient echo sequence (TR / TI / TE = 2300/900 /2.9 ms)
  3. an analysis of the anatomic connectivity of the patient's brain assessed using a 1.5mm isotopic DTI with a high number of directions (HARDI / 65 directions / b=1500s/mm2).
  4. An evaluation of neuronal dysfunction using MR Spectroscopy. Spectroscopic data will be collected using a 2D CSI laser with a short TE technique.
  5. Magnetization transfer imaging providing information about integrity of membranes.

SUMMARY:
To assess the neurocognitive outcomes in patients treated with chemotherapy for a malignant bone tumor during childhood and adolescence and the factors associated with neurocognitive impairment and/or complaints

ELIGIBILITY:
Inclusion Criteria:

For study OSE A and B

* Patients treated for a bone sarcoma: Ewing or osteosarcoma
* Age under 19 years at initial diagnosis
* Treated in the Pediatric Oncology Department of Gustave

For patients diagnosed between 01.01.2001 and 31.12.2010: patients alive in complete remission at least 5 years after diagnosis

* Treated with at least one course of HDMTX for osteosarcoma
* Treated without HDMTX for Ewing sarcoma
* Time interval between the end of treatment and inclusion >10 y
* Age > 21 y at inclusion
* Patients with informed consent signed
* Patient under guardianship
* Affiliated to French health insurance or beneficiary of the same or equivalent

For study OSE- B only:

* Treated with at least 8 courses of HDMTX for osteosarcoma
* Treated without HDMTX for Ewing sarcoma
* Patients with Ewing sarcoma will have to be matched with osteosarcoma patients according to age at the time of treatment, sex, and duration of follow-up
* School level equivalent of at least the end of primary school

Exclusion Criteria:

For study OSE A and B

* Brain radiotherapy
* Previous relapse except those treated by local treatment without any chemotherapy
* Second malignancy treated with chemotherapy
* High dose chemotherapy with stem cell support
* Non-French speaking patients
* Pregnant and breastfeeding women

For study OSE- B only:

- Patient deprived of his liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
scores obtained in FactCOG as a whole and in each subscale | 3 years
  Primary analysis will be performed on all patients included in the study, including history of Ewing (treated without HDMTX) and osteosarcoma (treated with HDMTX). This population is the main analysis population of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France